CLINICAL TRIAL: NCT01108458
Title: A Phase 2 Study of Pertuzumab and Erlotinib for Refractory Pancreatic Adenocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Extreme toxicity of Pertuzumab and Erlotinib combination
Sponsor: George Albert Fisher (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, George Albert Fisher, Associate Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-18227; SU-03082010-5163 (Other: Stanford University); PANC0010 (Other: OnCore)
Record Dates: First submitted 2010-04-20; First posted 2010-04-22 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — pertuzumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pertuzumab plus Erlotinib Hydrochloride (Experimental): Pertuzumab 840 mg intravenous (IV) single loading dose followed by 420 mg IV every 3 weeks
  Erlotinib hydrochloride 150 mg/day by mouth
  Interventions: Drug: Pertuzumab; Drug: Erlotinib

INTERVENTIONS:
Drug: Pertuzumab — iv, 840 mg, 420 mg
  Other Names: 2C4; Omnitarg
Drug: Erlotinib — PO, 150 mg
  Other Names: Erlotinib hydrochloride; Tarceva

SUMMARY:
A phase 2 study combining pertuzumab with erlotinib for patients with gemcitabine refractory pancreatic adenocarcinoma

DETAILED DESCRIPTION:
A single-institution, single-arm phase 2 study investigating pertuzumab and erlotinib as a palliative regimen in the treatment of locally-advanced or metastatic pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

3.1 Inclusion Criteria

3.1.1 Histologically-confirmed pancreatic adenocarcinoma

3.1.2 One or more locally-advanced or metastatic lesions measurable in at least one dimension by modified RECIST criteria (v1.1)^13 within 4 weeks prior to entry of study

3.1.3 Prior therapy (1 or more):

3.1.3.1 Disease progression following therapy with gemcitabine

3.1.3.2 Intolerance to gemcitabine

3.1.3.3 Disease recurrence within 12 months following adjuvant gemcitabine

3.1.4 Age >= 18

3.1.5 ECOG performance status 0-2

3.1.6 Laboratory values <= 2 weeks prior to enrollment:

* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (>= 1500/mm^3)
* Platelets (Plt) >= 100,000/mm^3
* Hemoglobin (Hgb) >= 9 g/dL
* Serum creatinine <= 1.5 x ULN
* Serum bilirubin <= 1.5 x ULN (<= 3.0 x ULN if liver metastases present)
* Aspartate aminotransferase (AST/SGOT), alanine aminotransferase (ALT/SGPT) <= 3.0 x ULN. (<= 5.0 x ULN if liver metastases present). ERCP or percutaneous stenting may be used to normalize the liver function tests

3.1.7 Echocardiogram or MUGA scan demonstrating LVEF >= 50% within 4 weeks of trial entry

3.1.8 Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

3.2 Disease-Specific Exclusion Criteria

3.2.1 Prior therapy with EGFR-targeted agents

3.2.2 If history of other primary cancer, subject will be eligible only if she or he has:

* Curatively resected non-melanomatous skin cancer
* Curatively treated cervical carcinoma in situ
* Other primary solid tumor curatively treated with no known active disease present and no treatment administered for the last 3 years

3.3 General Medical Exclusion Criteria

3.3.1 Subjects known to have chronic or active hepatitis B or C infection with impaired hepatic function (ineligible if AST and ALT > 3.0 x ULN).

3.3.2 History of any medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risks associated with study participation or study drug administration or may interfere with the conduct of the study or interpretation of study results

3.3.3 Male subject who is not willing to use adequate contraception upon enrollment into this study and for 6 months following the last dose of study agents

3.3.4 Female subject (of childbearing potential, post-menopausal for less than 6 months, not surgically sterilized, or not abstinent) who is not willing to use an oral, patch or implanted contraceptive, double-barrier birth control, or an IUD during the course of the study and for 6 months following the last dose of second-line treatment

3.3.5 Female subject who is breast-feeding or who has positive serum pregnancy test 72 hours prior to enrollment

3.3.6 Any of the following concurrent severe and/or uncontrolled medical conditions within 24 weeks of enrollment which could compromise participation in the study:

* Unstable angina pectoris
* Symptomatic congestive heart failure
* Myocardial infarction <= 6 months prior to registration and/or randomization
* Serious uncontrolled cardiac arrhythmia
* Uncontrolled diabetes
* Active or uncontrolled infection
* Interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung
* Chronic renal disease

3.3.7 Patients unwilling to or unable to comply with the protocol

3.3.8 Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech/Roche sponsored cancer study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-07; Primary Completion 2010-11 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Albert Fisher M.D. Ph.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pertuzumab Plus Erlotinib Hydrochloride: Pertuzumab 840 mg intravenous (IV) single loading dose followed by 420 mg IV every 3 weeks
  Erlotinib hydrochloride 150 mg/day by mouth
  Pertuzumab: iv, 840 mg, 420 mg
  Erlotinib: PO, 150 mg
Period: Overall Study
Arm/Group | Pertuzumab Plus Erlotinib Hydrochloride
Started | 1
Completed | 0
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pertuzumab Plus Erlotinib Hydrochloride
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Gender [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate by RECIST Criteria
Time Frame: CT imaging every 9 weeks while on protocol
Arm/Group | Pertuzumab Plus Erlotinib Hydrochloride
Number analyzed (Participants) | 0
Value | 0

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Disease status evaluated by computed tomography (CT) scan and progression-free survival assessed per RECIST criteria.
  Tumor response was assessed by the IRF according to RECIST v1.1. CR was defined as disappearance of all target and non-target lesions and (if applicable) normalization of tumor marker levels. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 millimeters (mm). PR was defined as greater than or equal to (≥) 30 percent (%) decrease in sum of longest diameter (LD) of target lesions in reference to Baseline sum LD. Response was to be confirmed ≥4 weeks after the initial assessment of CR or PR. The percentage of participants with a confirmed objective response of CR or PR was reported.
Time Frame: 9 weeks
Arm/Group | Pertuzumab Plus Erlotinib Hydrochloride
Number analyzed (Participants) | 0
Value | 0

3. Secondary Outcome: Overall Survival (OS)
Time Frame: 1 year
Arm/Group | Pertuzumab Plus Erlotinib Hydrochloride
Number analyzed (Participants) | 0
Value | 0

4. Secondary Outcome: Quality of Life (QoL)
Description: Quality of life as assessed by EORTC QLQ-C30 questionnaire
Time Frame: 3 weeks
Arm/Group | Pertuzumab Plus Erlotinib Hydrochloride
Number analyzed (Participants) | 0
Value | 0

5. Secondary Outcome: No. of Events of Drug-related Toxicity
Description: Number of incidences of serious and non-serious drug-related adverse events
Time Frame: 3 weeks
Measure: Number; unit: Drug-related adverse events
Arm/Group | Pertuzumab Plus Erlotinib Hydrochloride
Number analyzed (Participants) | 1
Drug-related adverse events | 3

6. Secondary Outcome: Proportion of Participants With 50% Decrease in Tumor Marker
Description: Change in tumor marker CA19-9, assessed as a 50% decrease from baseline
Time Frame: 3 weeks
Arm/Group | Pertuzumab Plus Erlotinib Hydrochloride
Number analyzed (Participants) | 0
Value | 0

ADVERSE EVENTS:
Arm/Group | Pertuzumab Plus Erlotinib Hydrochloride
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pertuzumab Plus Erlotinib Hydrochloride (N=1)
Fatigue (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No